CLINICAL TRIAL: NCT06337396
Title: Omic Approaches to Characterize the Functional and Phenotypic Consequences of Rare Structural Genomic Variants in Neurodevelopmental Disabilities and Congenital Anomalies
Brief Title: Omic Approaches to Neurodevelopmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1001
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Neurodevelopmental Disorders
Keywords: whole genome sequencing; transcriptome analysis; genotype phenotype; structural variants
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Transcriptome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Whole Genome Sequencing (WGS) and transcriptome analysis (Experimental): to investigate by WGS analysis the genome of selected patients with a detailed clinical characterization. WGS will be also performed on the DNA of the parent from which originated the CNV to look for any potential genomic signatures predisposing to the rearrangement detected in his/her son/daughter.
  to investigate the expression profiles of structural variants by transcriptome analysis
  Interventions: Diagnostic Test: WGS and transcriptome analysis

INTERVENTIONS:
Diagnostic Test: WGS and transcriptome analysis — In light of the inconsistencies between the CNV and the phenotypic outcome, we expect that WGS analysis will reveal that part of these CNVs have a more complex structure than the one disentangled by CMA and FISH. We hypothesize that CNV should reflect a perturbed genome folding configuration at several hierarchical levels of chromatin organization, such as disruption of TADs boundaries. To investigate this aspect, we plan to examine expression profiles of immortalized lymphoblastoid B-cell lines (LBLs) derived from normal controls and patients. We expect to find a subset of down- or up-regulated genes located inside the rearranged region which in turn may alter the expression of other genes, possibly leading to perturbation of disease-related pathways

SUMMARY:
to bridge the gap between the molecular structure of CNV and the effect on the phenotype, considering NDDs as complex diseases, as they are a consequence of the imbalance in several dosage-sensitive genes, we might try to approach them through different --omics investigations (genomics, epigenomics, transcriptomics) according to the emerging field of network medicine. This holistic can provide valuable insight into understanding peculiar molecular mechanisms and unsuspected molecular interactions that contribute to the pathogenesis of the condition and possibly pave the way for uncovering new drug strategies that even if they do not heal the patient may improve his performance and the social interaction

ELIGIBILITY:
Inclusion Criteria:

Patients with neurodevelopmental disorders carrying a genomic rearrangement identified through chromosomal microarray analysis (CMA)

Exclusion Criteria:

NA

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of likely pathogenic structural variants | once at recruitment
  Number of likely pathogenic structural variants found by whole genome sequencing and transcriptome analysis.
Number of patients for whom a genotype-phenotype correlation is found | once at recruitment
  Number of patients for whom a genotype-phenotype correlation is found based on results of whole genome sequencing and transcriptome analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No